CLINICAL TRIAL: NCT00131313
Title: A Multicenter, Open-Label Study of Nipent, Cytoxan and Rituxan in Patients With Previously Untreated or Treated Chronic Lymphocytic Leukemia.
Brief Title: Efficacy and Safety of Nipent, Cytoxan and Rituxan in the Treatment of Chronic Lymphocytic Leukemia.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Valley Hematology and Oncology Medical Group (Other)
Collaborators: Mena, Raul, M.D. (Individual); Pharmatech Oncology (Industry); Astex Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POI-02818; NIP-02-005
Record Dates: First submitted 2005-08-16; First posted 2005-08-18 (Estimated); Last update posted 2005-08-18 (Estimated); Status verified 2005-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Leukemia; Cancer; Nipent; Rituxan; Cytoxan
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia; Neoplasms | interventions — Pentostatin; Cyclophosphamide; Rituximab

INTERVENTIONS:
Drug: Nipent, Cytoxan, Rituxan

SUMMARY:
This research study measures the safety and efficacy of the combination of three drugs that are approved, Nipent, Rituxan and Cytoxan in the treatment of Chronic Lymphocytic Leukemia (CLL). These drugs are being given together for investigational purposes as the specific combination of these three drugs has not been approved for treatment of CLL by the FDA.

DETAILED DESCRIPTION:
Chronic Lymphocytic Leukemia (CLL) is the most common form of adult leukemia in the U.S. Recent experience with Nipent in conjunction with Rituxan has shown that this combination is well tolerated and is clinically promising. It is expected that the addition of Cytoxan in patients with previously untreated CLL and patients who have relapsed or failed prior therapy may benefit from combined therapy using Nipent, Cytoxan and Rituxan. It is unknown how the addition of Cytoxan will affect the toxicity profile of the Rituxan and Nipent regimen, however, patients will be monitored for toxicities. It is expected that bone marrow toxicities will not increase to unreasonable levels.

The primary objective of the study is to determine the overall efficacy response rate following treatment with Nipent, Cytoxan and Rituxan of patients with previously untreated or treated CLL. The secondary objectives of the study are to determine the duration of response, time to progression, time to treatment failure and to evaluate the toxicity of this combination of drugs and the incidence and severity of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Stage II, III or IV Chronic Lymphocytic Leukemia
* Disease requires chemotherapeutic treatment
* CT or MRI scan confirming measurable tumor size
* Documentation of CD markers
* Up to one prior treatment regimen
* Expected survival greater than 6 months
* ECOG performance status of 0-2
* Adequate renal, bone marrow and liver functions
* Negative pregnancy test (females of childbearing potential)
* Must agree to use acceptable birth control, if fertile
* Must complete Informed Consent
* No heart disease and must have adequate cardiac function
* Must test negative for viral Hepatitis B and C

Exclusion Criteria:

* More than one prior treatment for Chronic Lymphocytic Leukemia
* Known sensitivity to Nipent, Rituxan or Cytoxan or any component of these drugs
* Known HIV or AIDS illness
* Thyroid disease requiring medication
* History of any malignancy that could affect the diagnosis or assessment of the study treatment
* Pregnancy or breast feeding
* Evidence of Hepatitis B or C infection
* Inability to comply with the requirements of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180
Dates: Start 2003-01; Study Completion 2009-04

PRIMARY OUTCOMES:
Efficacy response rate

SECONDARY OUTCOMES:
Time to progression
Time to treatment failure
Toxicity
Incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Raul Mena, MD, Principal Investigator — East Valley Hematology and Oncology Group
Locations (52):
- United States (52):
  - Northwest Alabama Cancer Center, PC, Muscle Shoals, Alabama
  - East Valley Hematology and Oncology Medical Group, Burbank, California
  - Bay Area Cancer Research Group, Concord, California
  - Lalita Pandit, MD, Inc., Fountain Valley, California
  - Pacific Coast Hematology/Oncology Medical Group, Inc., Fountain Valley, California
  - Robert A. Moss, M.D. FACP, Inc., Fountain Valley, California
  - Metropolitan Hematology Oncology Medical Group, Los Angeles, California
  - North County Oncology, Oceanside, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Cancer and Blood Institute Medical Group, Rancho Mirage, California
  - St. Teresa Comprehensive Cancer Center, Stockton, California
  - Medical Group of North County, Vista, California
  - The Oncology Clinic, PC, Colorado Springs, Colorado
  - Mile High Oncology, Denver, Colorado
  - Palm Beach Institute of Hematology and Oncology, Boynton Beach, Florida
  - Integrated Community Oncology Network, Jacksonville, Florida
  - Osceola Cancer Center, Kissimmee, Florida
  - Pasco Hernando Oncology Associates, PA, New Port Richey, Florida
  - Pasco Pinellas Cancer Center, New Port Richey, Florida
  - Augusta Oncology Associates, PC, Augusta, Georgia
  - Spalding Oncology Services, Griffin, Georgia
  - St Luke's Mountain States Tumor Institute, Boise, Idaho
  - Oncology Hematology Assoc. of Northern Illinois, Gurnee, Illinois
  - Indiana Oncology Hematology Consultants, Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Cancer Care Center, New Albany, Indiana
  - Kentucky Cancer Clinic, Hazard, Kentucky
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Chesapeake Oncology Hematology Associates, Baltimore, Maryland
  - Auerbach Hematology Oncology Associates, Inc., Baltimore, Maryland
  - Genesee Cancer & Blood Disease Treatment Center, PC, Flint, Michigan
  - West Michigan Regional Cancer & Blood Center, Free Soil, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Branson Oncology Clinic, Branson, Missouri
  - St. Louis Hematology Oncology Specialists, Inc., St Louis, Missouri
  - Sierra Nevada Oncology Care, Carson City, Nevada
  - Nevada Cancer Center, Las Vegas, Nevada
  - The Center for Cancer and Hematologic Disease, Cherry Hill, New Jersey
  - Ellioth Fishkin, MD, Elizabeth, New Jersey
  - Westchester Hematology Oncology Associates, Mount Kisco, New York
  - Mid Dakota Clinic/Odyssey Research, Bismarck, North Dakota
  - Summa Health System Hospitals, Akron, Ohio
  - Nashat Y. Gabrail, MD, Inc., Canton, Ohio
  - Sambandam and Joseph Associates, Inc, Cranston, Rhode Island
  - Charleston Hematology Oncology, PA, Charleston, South Carolina
  - South Carolina Oncology Associates, Columbia, South Carolina
  - The Family Cancer Center, Collierville, Tennessee
  - C. Michael Jones, MD, PC, Germantown, Tennessee
  - JPS Center for Cancer Care, Fort Worth, Texas
  - Cache Valley Cancer Treatment & Research Clinic, Inc., Logan, Utah
  - Cancer Outreach Associates, PC, Abingdon, Virginia
  - Virginia Oncology Care, PC, Richlands, Virginia

REFERENCES:
- See also: Pharmatech - The Research Link website — http://www.pharmatech.com/